CLINICAL TRIAL: NCT05811832
Title: Evaluation of Balance, Physical Activity, Functional Capacity and Activities of Daily Living in Frail Elderly Individuals with COPD
Brief Title: Evaluation in Elderly Individuals with Chronic Obstructive Pulmonary Disease(COPD)
Status: Completed | Type: Observational
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Meral SERTEL, associate professor, Kırıkkale University
Other Study IDs: KirikkaleUniversity771
Record Dates: First submitted 2023-03-29; First posted 2023-04-13 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-04

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease)
Keywords: COPD (Chronic Obstructive Pulmonary Disease); fragility; geriatric
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 8 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Fragile elderly individuals with COPD: Patient evaluation form and socio-demographic form of all individuals participating in the study.
  properties will be questioned.To assess pulmonary functions at the assessment stage for all individuals pulmonary function test,Modified Medical Questionnaire to assess dyspnea research Council, to assess health-related quality of life, Saint George Respiratory Two Minute Walk Test to assess exercise capacity, frailty Frail fragility scale to detect fragility, Prisma-7 Vulnerability scale to assess fragility The scale is Pase to assess physical activity, Berg balance to assess balance. scale, digital hand dynamometer to evaluate quadriceps muscle strength, hand grip strength hand dynamometer to assess fatigue levels Fatigue Severity Scale will be used.
  Interventions: Other: Evaluation
- Non-fragile elderly individuals with COPD: Patient evaluation form and socio-demographic form of all individuals participating in the study.
  properties will be questioned.To assess pulmonary functions at the assessment stage for all individuals pulmonary function test,Modified Medical Questionnaire to assess dyspnea research Council, to assess health-related quality of life, Saint George Respiratory Two Minute Walk Test to assess exercise capacity, frailty Frail fragility scale to detect fragility, Prisma-7 Vulnerability scale to assess fragility The scale is Pase to assess physical activity, Berg balance to assess balance. scale, digital hand dynamometer to evaluate quadriceps muscle strength, hand grip strength hand dynamometer to assess fatigue levels Fatigue Severity Scale will be used.
  Interventions: Other: Evaluation

INTERVENTIONS:
Other: Evaluation — Modified Medical research Council , Saint George Respiratory Two Minute Walk Test,Frail fragility scale ,Prisma-7 Vulnerability scale,Pase,Berg balance scale,manual muscle test,quadriceps muscle strength, hand dynamometer,Fatigue Severity Scale

SUMMARY:
This study is conducted on the evaluation of balance, physical activity, functional capacity and activities of daily living in frail elderly individuals with COPD.

DETAILED DESCRIPTION:
Patient evaluation form and socio-demographic form of all individuals participating in the study. Characteristics will be questioned: Name-surname, address, telephone, age, gender, weight, height, body mass index, occupation, marital status, social security, any systemic other than COPD whether he has a disease, whether he has social security, whether he smokes, It will be questioned whether there is any other COPD patient in the family and whether there is pain. To assess pulmonary functions at the assessment stage for all individuals pulmonary function test to evaluate dyspnea Modified Medical Saint George Respiratory Research Council to assess health-related quality of life Two Minute Walk Test to assess exercise capacity, frailty Frail fragility scale to detect frailty, Prisma-7 Vulnerability scale to assess fragility The scale was Pase to assess physical activity, Berg Balance to assess balance scale, digital hand dynamometer to assess quadriceps muscle strength, hand grip hand dynamometer to assess strength, fatigue levels Fatigue Severity Scale will be used to evaluate.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with COPD according to the Gold criteria
* Be over 65 years old
* Volunteering to participate in the study
* Not having mental and communication problems that prevent filling out the questionnaires to be used in the research.
* Not having an attack in the last 2 months

Exclusion Criteria:

* Being in a COPD exacerbation process
* Having been diagnosed with a physical and mental illness
* Having unstable COPD
* Unstabile angina, previous Myocardial Infractus, uncontrolled hypertension, cancer, with functional limitations concomitant neurological or musculoskeletal disorders
* Currently addicted to alcohol or drugs
* Having severe vision and hearing problems
* Have had major surgery in the last few months
* History of recurrent significant clinical infection

Ages: 65 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly individuals aged 65-84 years diagnosed with COPD who are frail or non-fragile.
Sampling Method: Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Berg balance scale(BDO) | eight months
  The Berg balance scale (BDO) is a scale with 14 instructions and a score of 0-4 for each instruction by observing the patient's performance. 0 points are given when the patient is unable to perform the activity at all, while 4 points are given when the patient completes the activity independently. The highest score is 56, with 0-20 points indicating a balance disorder, 21-40 points indicating the presence of an acceptable balance, and 41-56 points indicating the presence of a good balance.
Two-minute walk Test | eight months
  It is recommended that the area where the test will be performed is a corridor with a flat and hard floor of 30 meters long. The goal is to walk the maximum distance he can walk in 2 minutes if he has a helper device he uses. If you have shortness of breath or fatigue, you are told to slow down and stop and then start again when you feel ready.
Physical activity scale for the elderly (PASE) | eight months
  The survey assesses the physical activity of older individuals over the past week and includes components of leisure, housework, and work-related physical activity. Never, rarely (1-2 days/week), sometimes (3-4 days/week) and often (5-7 days/week), while the duration of activities is classified as: Less than 1 hours, 1-2 hours to 2-4 hours and more than 4 hours.
Saint George Respiratory Survey | eight months
  A test that assesses health-related quality of life specific to individuals with respiratory diseases. questions 50 items divided into 3 areas: symptoms (8 items), activities (16 items), effects of the disease (26 items). The 3 sections of the test are scored separately and the total score is calculated. The scores vary from 0-100-0. A score of zero indicates normal and a score of 100 indicates the worst state of health.
Modified Medical Research Council scale(MMRC) | eight months
  The MMRC (modified Medical Research Council scale) is a scale scored between 0 and 4 based on various factors that produce a dyspnea sensation. Zero points only shorten my breath during heavy exercise; 4 points I can't leave the house because of my shortness of breath or I have shortness of breath while getting dressed and undressed
Frail fragility scale | eight months
  Proven to be an effective method of vulnerability detection. The patient's fatigue status, resistance, mobility, weight loss and other diseases were questioned and allowed to evaluate. The FRAIL scale, which consists of 5 items, scores 0 1-2 or 1 based on the patients' response and is evaluated as non-frail, 0 points pre-frail and >2 points fragile.

SECONDARY OUTCOMES:
Breathing function test | eight months
  Spirometry shows the maximum volume of air expelled by the challenging expiration (challenging vital capacity, FVC) from the maximum inspiration point and the volume of air expelled in the first second of this manoeuvre (1. The challenging expiration volume per second, FEV 1) should be measured and these two measurement ratios (FEV 1/FVC) should be calculated. Patients with COPD typically have both FEV 1 and FVC low. When FEV 1/FVC < 70%, the postbronchodilator indicates the presence of a non-fully reversible airflow limitation when FEV 1 < 80% of what is expected.
Prisma-7 Vulnerability scale | eight months
  The PRISMA-7 vulnerability scale is a seven-question survey recommended by the British Geriatric Association as a first-degree screening test. The questions are answered in a yes/no way.
hand dynamometer | eight months
  During the test, the patient sits in a sitting position in shoulder adduction, elbow in 90° flexion, forearm in neutral position, and measurements are performed three repetitions for the right and left sides. It is recorded in kg or pounds as a unit. The norm values for the measurement are 47-40 kg for men aged 20-69 years (2 kg less for the left hand) and 30-24 kg for women (1,5-2 kg less for the left hand).
digital hand dynamometer | eight months
  For quadriceps strength measurement, the test is started when elderly people sit on a flat surface with their hips and knees in 90° flexion and feet in a free, unsupported position. During the test, the "make test" technique, which requires isometric contraction, is applied. All measurements are taken by the same researcher twice from both legs of the participants with the same hand.
Fatigue Severity Scale | eight months
  Evaluates fatigue severity with 9 questions and scores are taken from 9 to 63 on the scale. Each question is scored between 0 (I do not agree at all) and 7 (I totally agree). A high score indicates increased fatigue intensity.

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin Köse, Principal Investigator — Master of Science student; Döndü Nur Keskin, Principal Investigator — Master of Science student; İlayda Karabayır, Principal Investigator — Master of Science student; Meral Sertel, Study Director — Associate professor lecturer; Selma Demir, Principal Investigator — Specialist doctor
Locations (1):
- Kirikkale High Specialization Hospital, Kırıkkale, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No